CLINICAL TRIAL: NCT07240480
Title: Validation of the Turkish Version of the DDIVAT Visual Acuity Measuring Device in a Turkish-speaking Population
Brief Title: Assessing the Turkish DDIVAT for Visual Acuity Measurement
Status: Not yet recruiting | Type: Observational
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Hande Guclu, Department Head - Ophthalmology (Trakya Univ.)-Principal Investigator, Trakya University
Other Study IDs: Turkish DDIVAT TrakyaUni
Record Dates: First submitted 2025-11-16; First posted 2025-11-21 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Visual Acuity; Refractive Errors; Myopia; Hyperopia; Astigmatism
Keywords: Visual Acuity; Refractive Errors
MeSH Terms: conditions — Refractive Errors; Myopia; Hyperopia; Astigmatism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants Undergoing Visual Acuity Testing: All enrolled participants (n = 200) will complete two visual acuity measurements during a single visit: one using the DDIVAT (Digital Device Independent Visual Acuity Test) Turkish version and one using the standard Snellen chart. The study compares the agreement and test-retest reliability of these two methods. No intervention, medication, or treatment is applied.
  Interventions: Diagnostic Test: DDIVAT Visual Acuity Test (Turkish Version)

INTERVENTIONS:
Diagnostic Test: DDIVAT Visual Acuity Test (Turkish Version) — Participants' visual acuity will be measured using the Turkish version of the DDIVAT digital visual acuity device and compared with Snellen chart results. No treatment or invasive procedure will be performed.

SUMMARY:
The goal of this observational methodological study is to validate the Turkish version of the DDIVAT visual acuity measuring device in a Turkish-speaking adult population.

The main questions it aims to answer are:

Does the Turkish version of the DDIVAT provide reliable and valid visual acuity measurements in Turkish speakers?

Are the results of the DDIVAT comparable to those obtained with the standard Snellen chart used in clinical practice?

Researchers will compare DDIVAT visual acuity test results with Snellen chart results to see if both methods produce consistent measurements.

Participants will:

Be adults aged 18 years or older, including both patients and healthy volunteers.

Undergo visual acuity testing using the DDIVAT system displayed on a smart TV connected to the university server.

Have their visual acuity re-measured using the standard Snellen optotype under the same conditions.

No medication or invasive procedure will be used. The study carries no risk to participants.

DETAILED DESCRIPTION:
This study is a non-interventional, observational methodological validation study designed to evaluate the validity and reliability of the Turkish version of the DDIVAT (Digital Distance Interactive Visual Acuity Test) in a Turkish-speaking population.

The DDIVAT visual acuity test was originally developed and validated at Democritus University of Thrace (Greece) and has been approved by the National Medicines Organization as a Class I medical device. The current study aims to determine whether the Turkish-translated version of this visual acuity measurement tool performs consistently and accurately among Turkish-speaking participants.

Visual acuity is one of the most fundamental components of a comprehensive ophthalmological examination. It measures the clarity or sharpness of vision, which can be influenced by refractive errors and a variety of ocular diseases. Accurate and accessible tools for measuring visual acuity are therefore essential in both clinical and research settings.

In this study, 200 adult participants (aged 18 years and older) will be recruited from Trakya University Hospital, Department of Ophthalmology (Edirne, Türkiye). The study population will include both healthy volunteers and patients presenting to the ophthalmology clinic.

Each participant will undergo two visual acuity measurements under standardized conditions:

DDIVAT visual acuity test (Turkish version), administered via a smart TV connected to the university's secure server.

Snellen chart test, which represents the standard clinical practice currently used at Trakya University Hospital.

Measurements will be taken monocularly (each eye tested separately) while participants wear their current optical correction (e.g., eyeglasses or contact lenses).

The study will compare the two measurement methods to determine:

The level of agreement between DDIVAT and Snellen test results.

The test-retest reliability of the Turkish DDIVAT.

Since no medication, invasive procedure, or experimental intervention will be applied, the study poses no potential risk to participants. All procedures will comply with the Declaration of Helsinki, Good Clinical Practice (GCP) principles, and relevant data protection regulations.

Collected data will be stored anonymously and used solely for research purposes. The findings are expected to provide evidence supporting the use of DDIVAT as a reliable digital visual acuity tool for Turkish-speaking populations, enhancing accessibility and standardization of visual testing in both clinical and teleophthalmology contexts.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older

Turkish-speaking individuals able to understand the study purpose

Willingness to participate and provide written informed consent

Participants with or without refractive errors (e.g., myopia, hyperopia, astigmatism)

Exclusion Criteria:

* Age below 18 years

Individuals unable to complete visual acuity testing

Presence of severe ocular pathology (e.g., corneal opacity, retinal detachment) that prevents accurate measurement

Cognitive or communication difficulties preventing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Turkish-speaking adults (aged 18 and older), including both healthy volunteers and ophthalmology clinic patients, will be recruited from Trakya University Hospital, Department of Ophthalmology (Edirne, Türkiye).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Agreement between DDIVAT (Turkish version) and Snellen chart visual acuity measurements | During a single study visit (same day assessment)
  The primary outcome is to assess the level of agreement between visual acuity scores obtained using the Turkish version of the DDIVAT digital visual acuity device and those obtained using the standard Snellen chart. Statistical analysis will include correlation and Bland-Altman agreement methods to evaluate consistency and validity between the two testing methods.

CONTACTS AND LOCATIONS:
Overall Officials: Hande Güçlü, M.D., Prof. Dr., Principal Investigator — Trakya University Teaching and Research Hospital

IPD SHARING:
Plan to Share IPD: No
This is a minimal-risk, non-interventional validation study conducted at a single institution. The collected data will be anonymized and analyzed internally. Individual participant-level data will not be shared outside Trakya University Faculty of Medicine due to institutional data-protection policies.

REFERENCES:
- [Background] Posar A, Visconti P. Early Motor Impairment in Children with Autism Spectrum Disorder. Turk Arch Pediatr. 2021 Nov;56(6):646-647. doi: 10.5152/TurkArchPediatr.2021.21168. No abstract available. PMID 35110066
- [Background] Daiber HF, Gnugnoli DM. Visual Acuity. 2023 May 29. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK563298/ PMID 33085445
- See also: Official site of the DDIVAT (Digital Device Independent Visual Acuity Test) developed at Democritus University of Thrace, Greece. — http://ddivat.med.duth.gr/DDiVAT/welcome.html